CLINICAL TRIAL: NCT04345393
Title: Translating Scientific Evidence Into Practice Using Digital Medicine and Electronic Patient Reported Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: The Cleveland Clinic (Other); Northwestern University (Other); RxHealth (Unknown); University of California, Davis (Other)
Responsible Party: Principal Investigator, Bruce E. Sands, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: GCO 18-2481; STUDY-21-01875 (Other: Icahn School of Medicine at Mount Sinai); SSU00171350 (Other: Advarra)
Record Dates: First submitted 2020-03-20; First posted 2020-04-14 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: IBD; Treat to target; Digital transformation network; Social determinants of health; e-PRO
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — dystrobrevin

STUDY DESIGN:
Intervention Model Description: 1. Smartphone, and inform them about the DTN program through a description and embedded video.
  2. Including SDH, behavioral health, lack of knowledge of quality metrics, or lack of Smartphone access or connectivity.
  3. The IBD home or to IBDTx care pathways. RxUniverse platform allows the creation of adaptive pathways based on feedback loops that provide relevant on-demand resources based on patient care touch-points.
  4. Digitally enabled population, or an Interactive Voice Response [IVR] for those who are not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Transformation Network (DTN) Program (Experimental): IBD patients at the 3 sites will be sent a message to their Smartphone
  Interventions: Behavioral: Digital Transformation Network (DTN) Program
- Control Arm (Active Comparator): Patients will enter the control group once they initially complete the ePRO and online assessment tools. They will remain in the control group, and then at set intervals each site will transition these patients into the DTN intervention arm.
  Interventions: Behavioral: Digital Transformation Network (DTN) Program

INTERVENTIONS:
Behavioral: Digital Transformation Network (DTN) Program — Patients will be screened based on ePRO and online assessment tool results to be identified to be eligible for enrollment into the DTN program. The results of ePROs and online assessments will be used to precision match patients to in-person care at the IBD home or to IBDTx care pathways. RxUniverse platform allows the creation of adaptive pathways based on feedback loops that provide relevant on-demand resources based on patient care touch-points. For example, a patient with mild depression or anxiety, maybe offered an online DTx and if not useful, link to telepsychiatry or in-person psychiatry consultation. Patients will transition into the intervention DTN arm at set intervals by site.

SUMMARY:
Delivery of healthcare has been traditionally limited to in-person visits or hospitalizations, while patients spend the majority of their time at home or work. Digital Medicine (e.g. apps, remote monitoring, telemedicine, patient reported outcomes) has the potential to bridge this gap, but the question remains as to how to translate it to mainstream practice while providing individualized recommendations to improve population health across organizations. Through the creation of a Digital Transformation Network (DTN) for Inflammatory Bowel Disease (IBD), the study team plans to reduce digital disparities and scientifically test the impact of these technologies in a clinical trial in three CTSA sites catering to diverse populations and communities.

DETAILED DESCRIPTION:
Delivery of healthcare has been traditionally limited to in-person office visits or hospitalizations, while patients spent the majority of their time at home or work. Digital Medicine (e.g. apps, remote monitoring, telemedicine, patient reported outcomes ePRO has the potential to bridge this gap, but it is unclear how to implement in a mainstream clinical practice that can lead to high-level patient and provider adoption. Through the creation of a Digital Transformation Network (DTN) for Inflammatory Bowel Disease (IBD), the study team plans to reduce digital disparities and scientifically address the evidence gap of digital health interventions across populations and communities.

AIM I. Unify existing digital assets (mobile app, ePROs, assessment for digital disparities and behavioral health, referral to IBD home and health education) into an IBD Digital Therapeutics Toolkit and integrate with EHRs at 3 CTSA hubs. Hypothesis: Integration with EHRs will lead to higher adoption by providers and limit disruption of workflow.

AIM II: Establish baseline levels of digital connectivity, disease control, quality of life and care metrics in cohorts at the three IBD centers. Hypothesis: A multipronged approach of assessment through text, phone, an app, and in-person will yield higher adoption.

AIM III. Implement and evaluate precision-matched interventions (digital skills, social determinants, behavioral health, monitoring through apps, and referral to interdisciplinary care) among 1500 patients with IBD using a stepped-wedge, cluster- randomized trial. Hypothesis: Medical homes supported by a unified platform will translate to sustainable improvement in population health outcomes. Analyze the Impact of DTN interventions. The primary outcome will be the improvement of the percentage of patients in DTN in disease control and decrease in urgent care utilization (emergency department visits and hospitalization days) across the three CTSA sites.

AIM IV. Support sustainability and dissemination across CTSA sites. Hypothesis: The patient- centric DTN will be sustainable through alignment with value-based healthcare.

Anticipated Impact: About 2 million Americans suffer from IBD and many more with chronic inflammatory diseases. The study team hopes that this study will help the study team build an evidence-based approach to determine whether digital medicine can engage a diverse group of patients and improve outcomes; and if yes, how it can be reproduced and replicated across different settings to address theT3 and T4 translational gaps.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed Inflammatory Bowel Disease (IBD) will be enrolled into DTN in stepped-wedge cluster randomized trial
* Age greater than or equal to 18 years
* Ability to speak or understand English or Spanish Language.

Exclusion Criteria:

- Condition or disease that, in the opinion of the investigators, may make it exceedingly difficult for the patient to use DTN, including, but not limited to, advanced dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants in Disease Control | 1 year after enrollment
  Number of participants in disease control. Disease control is defined by normalization of inflammatory markers and ePROs (PRO2<8 and PRO3<13). PRO2 measures stool frequency and bleeding while PRO3 measures the number of liquid or soft stools, abdominal pain and general well-being. Inflammatory markers including Erythrocyte Sedimentation Rate (ESR), C-Reactive Protein (CRP) and Fecal Calprotectin will be dichotomized using cut-offs of <30mm/hr, <5mg/L and <50 μg/g respectively for normal values.
Change in Number of Unplanned Acute Care | baseline
  Change in number of unplanned acute care 1 year after enrollment as compared to baseline. Unplanned acute care is defined as the number of ED visits and hospitalizations days 12 months before the intervention and the last 12 months of DTN intervention.

SECONDARY OUTCOMES:
Northstar Digital Literacy Assessment | 1 year after enrollment
  Digital skills and connectivity will be assessed using the Northstar digital literacy assessment. A 17-item rating scale, with full score from 0 to 100, with score 85% or above achieve a passing score.
Digital Disparities Module | 1 year after enrollment
  The digital disparities module is still in development through SBIR. The digital disparities module will assess the impact of digital disparities module in improving digital skills and access to Internet using previously developed digital disparities assessment instrument. The scale for the digital disparities assessment full scale from 0 - 100 where a higher score indicates the patient has a higher level of disparity in digital connectivity, digital skills and digital usage.
Overall Health Numeric Rating Scale [OHNRS] | 1 year after enrollment
  Overall Health Numeric Rating Scale (OHNRS) - Full scale from 0 to 10, higher score indicates worse health outcomes
PROMIS Global scales | 1 year after enrollment
  PROMIS Global scales is a 14-item measure that is part of the PROMIS Social Function. The measure refers to social roles, such as work and family responsibilities, and more discretionary social activities, such as leisure activity and relationships with friends. standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Patient Health Questionnaire (PHQ-4) | 1 year after enrollment
  The Patient Health Questionnaire (PHQ)-4 s a 4 item inventory. Anxiety subscale from 0-6, depression subscale from 0-6, with full scale from 0-12, higher score indicates more symptoms.
Patient Health Questionnaire (PHQ-9) | 1 year after enrollment
  The Questionnaire Type 9 for Depression (PHQ-9) is a self-administered instrument. Full scale from 0-27, with higher score indicating more severe symptoms. As needed.
Generalized Anxiety Disorder scale (GAD-7) | 1 year after enrollment
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire. Full scale from 0-21, with higher score indicating more symptoms. As needed.
Number of participants with improvement in mucosal healing | 1 year after enrollment
  This will be defined as the absence of inflammation on endoscopy (scoring systems) or imaging notes collected from EHR.
Visual Analog Scale (VAS) | 1 year after enrollment
  The Visual Analog Scale (VAS) will be used to assess medication adherence using <80% cut-off to designate non-adherence. Full Scale from 0 to 100 with higher score indicating more adherence.
Proportion of patients meeting eligible quality metrics | 1 year after enrollment
  Proportion of patients meeting eligible quality metrics confirmed through EHR. Composite score of metrics for skin care protection, flu vaccination, smoking cessation advice, pneumonia vaccination, bone density test, hepatitis B screen steroid sparing medication, TB test and TPMT test
System Usability Scale (SUS) | 1 year after enrollment
  The system usability scale (SUS) is a 10-item Likert scale questionnaire. The range of scores is from 0 - 100 where a SUS score above 68 is considered average.
Net Promoter Score | 1 year after enrollment
  The Net Promoter is a 10 point scale and the full score ranges from -100 to 100 where a higher score translates to higher satisfaction with a product.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Sands, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - University of California, Davis, Davis, California
  - RxHealth, Secaucus, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391

DOCUMENTS (1):
  • Informed Consent Form (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT04345393/ICF_000.pdf